CLINICAL TRIAL: NCT01387607
Title: A 14-week, Randomized, Double-blind Placebo-controlled Study For Pregabalin In Subjects With Fibromyalgia
Brief Title: A Study For Pregabalin In Patients With Fibromyalgia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer's Upjohn has merged with Mylan to form Viatris Inc. (Industry)
Responsible Party: Sponsor
Organization: Pfizer (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A0081241
Record Dates: First submitted 2011-06-30; First posted 2011-07-04 (Estimated); Results first posted 2018-07-30 (Actual); Last update posted 2021-01-28 (Actual); Status verified 2017-09

CONDITIONS: Fibromyalgia
Keywords: Pregabalin; fibromyalgia
MeSH Terms: conditions — Fibromyalgia | interventions — Pregabalin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pregabalin (Experimental)
  Interventions: Drug: pregabalin
- Placebo (Placebo Comparator): Matched placebo
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: pregabalin — Pregabalin capsule, 300-450mg/day, twice daily
  Arms: Pregabalin
Drug: placebo — Placebo, twice daily
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and tolerability of pregabalin compared with placebo for management of fibromyalgia in adults.

ELIGIBILITY:
Inclusion Criteria:

* Male or female patients, at least 18 years of age
* Meeting the ACR (America College of Rheumatology) criteria for fibromyalgia (ie, widespread pain present for at least 3 months, and pain in at least 11 of 18 specific tender point sites)
* At screening (V1) and randomization (V2), patients must have a score of no less than 40 mm on the Pain Visual Analog Scale (VAS)
* At randomization (V2), at least 4 pain diaries must be completed satisfactorily within the last 7 days and the average pain score must be no less than 4

Exclusion Criteria:

* Patients with no less than 30% decrease on the Pain Visual Analog Scale (VAS) at randomization (V2) as compared to screening (V1)
* Patients with other severe pain due to other conditions (eg, DPN or PHN) that may confound assessment or self-evaluation of the pain associated with fibromyalgia
* Patients with any widespread inflammatory musculoskeletal disorders, widespread rheumatic diseases other than fibromyalgia, active infections, or untreated endocrine disorders
* CLcr less than 60 mL/min (estimated from serum creatinine)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 343 (Actual)
Dates: Start 2012-02-06 (Actual); Primary Completion 2016-10-31 (Actual); Study Completion 2016-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (22):
- China (22):
  - Department of Rheumatism And Immunity, The First Affiliated Hospital of Bengbu Medical College, Bengbu, Anhui
  - Anhui Province Hospital, Hefei, Anhui
  - Beijing Chao-Yang Hospital, Capital Medical University, Beijing, Beijing Municipality
  - Southwest Hospital of the Third Military Medical University,PLA, Chongqing, Chongqing Municipality
  - Department of Neurology,General Hospital of Guangzhou Military Command of PLA, Guangzhou, Guangdong
  - Guangdong General Hospital, Guangzhou, Guangdong
  - Department of Neurology,The First Affiliated Hospital Of Guangzhou Medical University, Guangzhou, Guangdong
  - The Third Affiliated Hospital Of Sun Yat-sen University, Guangzhou, Guangdong
  - Rheumatology Department, The first Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Rheumatology Department, The second Affiliated Hospital of Harbin Medical University, Harbin, Heilongjiang
  - Xiangya Hospital of Centre-south University, Changsha, Kaifu District, Hunan
  - The Second Affiliated Hospital to Nanchang University, Nanchang, Jiangxi
  - Zhongshan Hospital Fudan University, Rheumatology Department, Shanghai, Shanghai Municipality
  - Xijing Hospital, The Fourth Military Medical University, Xi’an, Shanxi
  - Si Chuan Huaxi Hospital/Rheumatology Department, Chengdu, Sichuan
  - The First Affiliated Hospital of Kunming Medical University/ Rheumatology and Immunology Department, Kunming, Yunnan
  - The First Affiliated Hospital of Wenzhou Medical University/Neurology Department, Wenzhou, Zhejiang
  - China-Japan Friendship Hospital/Rheumatology Department, Beijing
  - Peking Union Medical College Hospital/Rheumatology Department, Beijing
  - PLA. The Military General Hospital of Beijing, Beijing
  - Rheumatology and Immunology Dept., Renji Hospital Shanghai Jiao Tong University School of Medicine, Shanghai
  - Rheumatology and Immunology Department, Shanghai Changzheng Hospital, Shanghai

REFERENCES:
- [Derived] Zhang X, Xu H, Zhang Z, Li Y, Pauer L, Liao S, Zhang F. Efficacy and Safety of Pregabalin for Fibromyalgia in a Population of Chinese Subjects. J Pain Res. 2021 Feb 25;14:537-548. doi: 10.2147/JPR.S281483. eCollection 2021. PMID 33658841
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0081241&StudyName=A%20Study%20For%20Pregabalin%20In%20Patients%20With%20Fibromyalgia%20

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: A total of 431 participants were screened and 343 of these were randomized. A total of 334 participants received the assigned study treatment.
Groups:
- Pregabalin: Pregabalin was administered orally, at a dose level of 75 mg (1 capsule) twice daily (BID) (Day 0 evening - Day 7 morning) and 150 mg (1 capsule) BID (Day 7 evening - Day 14 morning) in the titration phase.
  Pregabalin was then administered at a dose level of 150 mg (1 capsule) BID or 225 mg (2 capsules; 75 mg + 150 mg) BID in Day 14 evening and Weeks 3 - 14 during the fixed-dose phase. A 1-week taper off dose phase was in the following with pregabalin 150 mg or 225 mg administered in the morning and 75 mg administered in the evening.
- Placebo: Placebo matched to pregabalin 75 mg (1 capsule) was administered twice daily (BID) (Day 0 evening - Day 7 morning) and 150 mg (1 capsule) BID (Day 7 evening - Day 14 morning) in the titration phase. Placebo was then administered as matched to pregabalin 150 mg (1 capsule) BID or 225 mg (2 capsules; 75 mg + 150 mg) BID in Day 14 evening and Weeks 3 - 14 during the fixed-dose phase. A 1-week taper off dose phase was in the following with placebo matched to pregabalin 150 mg or 225 mg administered in the morning and 75 mg administered in the evening.
  Number of capsules taken daily with placebo matched the number taken for the assigned pregabalin dose level.
Period: Overall Study
Arm/Group | Pregabalin | Placebo
Started | 173 | 170
Received Treatment | 170 | 164
Completed | 122 | 125
Not Completed | 51 | 45
Not completed — Adverse Event | 23 | 11
Not completed — Lack of Efficacy | 8 | 6
Not completed — Lost to Follow-up | 2 | 1
Not completed — No longer meets eligibility criteria | 0 | 1
Not completed — Protocol Violation | 1 | 5
Not completed — Withdrawal by Subject | 13 | 14
Not completed — Other | 1 | 1
Not completed — Randomized, not treated | 3 | 6

BASELINE CHARACTERISTICS:
Population: The Full Analysis Set (FAS) was defined as all randomized participants who received at least 1 dose of study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Pregabalin | Placebo | Total
Number analyzed (Participants) | 170 | 164 | 334
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.5 (11.5) | 43.5 (10.6) | 44.0 (11.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 142 | 144 | 286
  Male | 28 | 20 | 48
Primary Diagnoses and Durations [Mean (Standard Deviation); unit: years]
  Fibromyalgia duration since onset of symptoms | 6.0 (7.0) | 5.6 (6.4) | 5.8 (6.7)
  Fibromyalgia duration since diagnosis | 0.3 (1.0) | 0.4 (1.2) | 0.3 (1.1)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Endpoint Mean Pain Score During the Double-blind Treatment Period at Week 14
Description: Assessment of mean pain score was based on participant's daily pain diary. The daily pain diary consisted of an 11-point numeric rating scale ranging from 0 (no pain) to 10 (worst possible pain). The participants rated their pain during the past 24 hours by choosing the appropriate number between 0 and 10. Self-assessment was performed daily at awakening. The endpoint mean pain score was defined as the mean of the Week 14 pain diary entries in the double-blind treatment phase. Baseline was defined as the mean of last 7 pain diary entries up to and including Day 1.
Time Frame: Baseline, Week 14
Population: The Full Analysis Set (FAS) was defined as all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 128 | 124
Units on a scale | -2.01 (0.148) | -1.28 (0.150)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0001, Mixed-effects model repeated measures — From a repeated measures analysis (MMRM) with treatment, pooled center, week, and treatment-by-week interaction as factors, and baseline value as covariate; Mean Difference (Final Values) = -0.730, 95% CI 2-sided [-1.10 to -0.36], Standard Error of Mean 0.1906

2. Secondary Outcome: Percentage of Participants Categorized by Each Patient Global Impression of Change (PGIC) Score at Week 14
Description: The Patient Global Impression of Change (PGIC) was a participant-rated instrument that measured change in participant's overall status on a scale ranging from 1 (very much improved) to 7 (very much worse), which was based on a validated scale, the Clinical Global Impression of Change (CGIC). Categories were defined based on the PGIC scores as followed: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse and 7 = very much worse.
Time Frame: Week 14
Population: The Full Analysis Set (FAS) was defined as all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 142 | 142
Percentage of participants
  Very much improved | 9.9 | 7.7
  Much improved | 25.4 | 19.7
  Minimally improved | 40.1 | 42.3
  No change | 17.6 | 24.6
  Minimally worse | 4.9 | 3.5
  Much worse | 2.1 | 2.1
  Very much worse | 0.0 | 0.0
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Statistical analysis performed for PGIC endpoint re-categorized into much/very much improved and other; Test type: Superiority or Other; p = 0.1397, Cochran-Mantel-Haenszel — Based on the combined categories from Cochran-Mantel-Haenszel test adjusted for pooled center; Odds Ratio (OR) = 1.4376, 95% CI 2-sided [0.8732 to 2.3667] — Overall odds ratio was calculated based on Mentel-Haenszel method as pregabalin versus placebo
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis performed for PGIC endpoint re-categorized into any improvement (participants who were very much improved or much improved or minimally improved) and other; Test type: Superiority or Other; p = 0.1510, Cochran-Mantel-Haenszel — Based on the combined categories from Cochran-Mantel-Haenszel test adjusted for pooled center; Odds Ratio (OR) = 1.4626, 95% CI 2-sided [0.8596 to 2.4886] — Overall odds ratio was calculated based on Mentel-Haenszel method as pregabalin versus placebo

3. Secondary Outcome: Change From Baseline in Fibromyalgia Impact Questionnaire (FIQ) Total Score at Week 14
Description: The Fibromyalgia Impact Questionnaire (FIQ) was a 20-item participant-reported outcome instrument designed to assess health status, progress, and outcomes in participants with fibromyalgia. It contained 10 subscales. There were 11 questions that are related specifically to physical functioning. The remaining items assessed pain, fatigue, stiffness, difficulty working, and symptoms of anxiousness and depression. Score range for each subscale was 0 to 10. The 10 subscales were combined to yield a total score with range from 0 to 100. The total score provided an estimation of fibromyalgia impact with higher scores indicating greater impairment.
Time Frame: Baseline, Week 14
Population: The Full Analysis Set (FAS) was defined as all randomized participants who received at least 1 dose of study medication. Last observation carried forward (LOCF) method was used.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 170 | 164
Units on a scale | -11.14 (1.343) | -8.15 (1.367)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0762, ANCOVA — From the analysis of covariate (ANCOVA) with treatment and pooled center as factors, and baseline value as covariate; Mean Difference (Final Values) = -2.990, 95% CI 2-sided [-6.30 to 0.32], Standard Error of Mean 1.6804

4. Secondary Outcome: Percentage of Participants With at Least 30% Reduction in Weekly Mean Pain Score From Baseline to Week 14
Description: Assessment of mean pain score was based on participant's daily pain diary. The daily pain diary consisted of an 11-point numeric rating scale ranging from 0 (no pain) to 10 (worst possible pain). The participants rated their pain during the past 24 hours by choosing the appropriate number between 0 and 10. Self-assessment was performed daily at awakening. Weekly mean pain score was calculated as mean value of the observations within the window for each week during the double-blind treatment phase. A participant with at least 30% reduction in weekly mean pain score from baseline to Week 14 was defined as a 30% responder.
Time Frame: Baseline, Week 14
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 162 | 159
Percentage of participants | 47.5 | 32.7
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0044, Cochran-Mantel-Haenszel — From Cochran-Mantel-Haenszel test comparing pregabalin to placebo adjusted for pooled center; Odds Ratio (OR) = 1.8924, 95% CI 2-sided [1.2007 to 2.9827] — Overall odds ratio was calculated based on Mantel-Haenszel method as pregabalin versus placebo

5. Secondary Outcome: Percentage of Participants With at Least 50% Reduction in Weekly Mean Pain Score From Baseline to Week 14
Description: Assessment of mean pain score was based on participant's daily pain diary. The daily pain diary consisted of an 11-point numeric rating scale ranging from 0 (no pain) to 10 (worst possible pain). The participants rated their pain during the past 24 hours by choosing the appropriate number between 0 and 10. Self-assessment was performed daily at awakening. Weekly mean pain score was calculated as mean value of the observations within the window for each week during the double-blind treatment phase. A participant with at least 50% reduction in weekly mean pain score from baseline to Week 14 was defined as a 50% responder.
Time Frame: Baseline, Week 14
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 162 | 159
Percentage of participants | 27.2 | 17.0
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0189, Cochran-Mantel-Haenszel — From Cochran-Mantel-Haenszel test comparing pregabalin to placebo adjusted for pooled center; Odds Ratio (OR) = 1.9683, 95% CI 2-sided [1.1151 to 3.4742] — Overall odds ratio was calculated based on Mantel-Haenszel method as pregabalin versus placebo

6. Secondary Outcome: Change From Baseline at Week 14 in Medical Outcome Study (MOS)-Sleep Scale - Sleep Disturbance Subscale Score
Description: The Medical Outcomes Study (MOS)-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assess key constructs of sleep. Instrument scoring yields 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. Range of scores represented for sleep disturbance was 0 to 100, with higher scores indicating more of the attribute.
Time Frame: Baseline, Week 14
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 169 | 164
Units on a scale | -11.45 (1.608) | -8.02 (1.636)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0900, ANCOVA — From the analysis of covariance (ANCOVA) with treatment and pooled center as factors and baseline value as covariate; Mean Difference (Final Values) = -3.427, 95% CI 2-sided [-7.39 to 0.54], Standard Error of Mean 2.0152

7. Secondary Outcome: Change From Baseline at Week 14 in Medical Outcome Study (MOS)-Sleep Scale - Snoring, Awaken Short of Breath and Sleep Adequacy Subscale Scores
Description: The Medical Outcomes Study (MOS)-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assess key constructs of sleep. Instrument scoring yields 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. Range of scores represented for snoring, awaken short of breath and sleep adequacy was 0 to 100, with higher scores indicating more of the attribute.
Time Frame: Baseline, Week 14
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 170 | 164
Units on a scale
  Snoring | 4.61 (1.748) | 2.08 (1.777)
  Awaken Short of Breath | -6.76 (1.809) | -4.41 (1.842)
  Sleep Adequacy | 14.23 (1.940) | 5.20 (1.990)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Statistical analysis for snoring; Test type: Superiority or Other; p = 0.2485, ANCOVA — From the analysis of covariance (ANCOVA) with treatment and pooled center as factors and baseline value as covariate; Mean Difference (Final Values) = 2.527, 95% CI 2-sided [-1.77 to 6.83], Standard Error of Mean 2.1858
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis for awaken short of breath; Test type: Superiority or Other; p = 0.2993, ANCOVA — From the analysis of covariance (ANCOVA) with treatment and pooled center as factors and baseline value as covariate; Mean Difference (Final Values) = -2.355, 95% CI 2-sided [-6.81 to 2.10], Standard Error of Mean 2.2650
Statistical Analysis 3: Comparison: Pregabalin vs Placebo; Statistical analysis for sleep adequacy; Test type: Superiority or Other; p = 0.0003, ANCOVA — From the analysis of covariance (ANCOVA) with treatment and pooled center as factors and baseline value as covariate; Mean Difference (Final Values) = 9.030, 95% CI 2-sided [4.21 to 13.85], Standard Error of Mean 2.4485

8. Secondary Outcome: Change From Baseline at Week 14 in Medical Outcome Study (MOS)-Sleep Scale - Quantity of Sleep and Somnolence Subscale Scores
Description: The Medical Outcomes Study (MOS)-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assess key constructs of sleep. Instrument scoring yields 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. Range of quantity of sleep parameter was 0 to 24 and somnolence was 0 to 100, with higher scores indicating more of the attribute.
Time Frame: Baseline, Week 14
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 170 | 163
Units on a scale
  Quantity of Sleep | 0.61 (0.089) | 0.32 (0.090)
  Somnolence | -1.29 (1.311) | -5.48 (1.337)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Statistical analysis for quantity of sleep; Test type: Superiority or Other; p = 0.0106, ANCOVA — From the analysis of covariance (ANCOVA) with treatment and pooled center as factors and baseline value as covariate; Mean Difference (Final Values) = 0.286, 95% CI 2-sided [0.07 to 0.51], Standard Error of Mean 0.1114
Statistical Analysis 2: Comparison: Pregabalin vs Placebo; Statistical analysis for somnolence; Test type: Superiority or Other; p = 0.0112, ANCOVA — From the analysis of covariance (ANCOVA) with treatment and pooled center as factors and baseline value as covariate; Mean Difference (Final Values) = 4.194, 95% CI 2-sided [0.96 to 7.43], Standard Error of Mean 1.6428

9. Secondary Outcome: Change From Baseline at Week 14 in Medical Outcome Study (MOS)-Sleep Scale - Sleep Problems Index Overall Score
Description: The Medical Outcomes Study (MOS)-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assess key constructs of sleep. Instrument scoring yields 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index. Range of sleep problem index overall score was 0 to 100, with higher scores indicating more of the attribute.
Time Frame: Baseline, Week 14
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 169 | 163
Units on a scale | -9.70 (1.307) | -6.64 (1.334)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0637, ANCOVA — From the analysis of covariance (ANCOVA) with treatment and pooled center as factors and baseline value as covariate; Mean Difference (Final Values) = -3.059, 95% CI 2-sided [-6.29 to 0.18], Standard Error of Mean 1.6438

10. Secondary Outcome: Percentage of Participants With Optimal Sleep at Week 14 in Medical Outcome Study (MOS)-Sleep Scale
Description: The Medical Outcomes Study (MOS)-Sleep Scale was a participant-rated questionnaire consisting of 12 items that assess key constructs of sleep. Instrument scoring yields 7 subscales (sleep disturbance, snoring, awaken short of breath or with a headache, quantity of sleep, optimal sleep, sleep adequacy, and somnolence) as well as a 9-item overall sleep problems index.
Time Frame: Baseline, Week 14
Population: as for outcome 3
Measure: Number; unit: Percentage of participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 170 | 163
Percentage of participants | 41.2 (41.2) | 43.6 (43.6)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.6767, Regression, Logistic — Logistic regression model includes treatment and pooled center as factors and baseline value as covariate; Odds Ratio (OR) = 1.12, 95% CI 2-sided [0.67 to 1.87]

11. Secondary Outcome: Change From Baseline in Mean Sleep Interference Score at Week 14
Description: The Daily Sleep Interference Scale was an 11-point numerical scale ranging from 0 (does not interfere with sleep) to 10 (completely interferes [unable to sleep due to pain]). Participants were asked to describe how their pain had interfered with their sleep during the past 24 hours by choosing the appropriate number between 0 and 10. Self-assessment was performed daily upon awakening. Baseline Mean Sleep Interference score was defined as the mean of all available last 7 sleep interference score diary entries up to and including Day 1.
Time Frame: Baseline, Week 14
Population: The Full Analysis Set (FAS) was defined as all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 128 | 124
Units on a scale | -1.88 (0.150) | -1.00 (0.153)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.882, 95% CI 2-sided [-1.26 to -0.50], Standard Error of Mean 0.1932

12. Secondary Outcome: Change From Baseline at Week 14 in Subjective Sleep Questionnaire (SSQ) - Subjective Wake After Sleep Onset (sWASO)
Description: The Subjective Sleep Questionnaire (SSQ) was included in the participant's diary and designed to capture subjective evaluation of sleep behavior in participants with disrupted sleep. It was administered to each participant approximately 30 - 60 minutes after arising each day in the morning. The Subjective Wake after Sleep Onset (sWASO) parameter subjectively estimated the total amount of time the participant was awake after initial sleep onset until final awakening. Baseline was defined as the mean of last 7 SSQ diary entries up to and including Day 1.
Time Frame: Baseline, Week 14
Population: The Full Analysis Set (FAS) was defined as all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 121 | 117
Minutes | -42.36 (5.920) | -25.19 (6.010)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0273, Mixed-effects model repeated measures — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -17.172, 95% CI 2-sided [-32.42 to -1.92], Standard Error of Mean 7.7785

13. Secondary Outcome: Change From Baseline at Week 14 in Subjective Sleep Questionnaire (SSQ) - Subjective Latency to Sleep Onset (sLSO)
Description: The Subjective Sleep Questionnaire (SSQ) was included in the participant's diary and designed to capture subjective evaluation of sleep behavior in participants with disrupted sleep. It was administered to each participant approximately 30 - 60 minutes after arising each day in the morning. The Subjective Latency to Sleep Onset (sLSO) parameter subjectively estimated the amount of time to fall asleep after lights out. Baseline was defined as the mean of last 7 SSQ diary entries up to and including Day 1.
Time Frame: Baseline, Week 14
Population: The Full Analysis Set (FAS) was defined as all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 124 | 122
Minutes | -0.26 (0.052) | -0.28 (0.053)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.8082, Mixed-effects model repeated measures — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.016, 95% CI 2-sided [-0.12 to 0.15], Standard Error of Mean 0.0677

14. Secondary Outcome: Change From Baseline at Week 14 in Subjective Sleep Questionnaire (SSQ) - Subjective Number of Awakenings After Sleep Onset (sNAASO)
Description: The Subjective Sleep Questionnaire (SSQ) was included in the participant's diary and designed to capture subjective evaluation of sleep behavior in participants with disrupted sleep. It was administered to each participant approximately 30 - 60 minutes after arising each day in the morning. The Subjective Number of Awakenings after Sleep Onset (sNAASO) parameter subjectively estimated the total number of times the participant awakened during the night until final awakening. Baseline was defined as the mean of last 7 SSQ diary entries up to and including Day 1.
Time Frame: Baseline, Week 14
Population: The Full Analysis Set (FAS) was defined as all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Awakenings
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 127 | 123
Awakenings | -0.95 (0.094) | -0.30 (0.095)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p < 0.0001, Mixed-effects model repeated measures — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = -0.655, 95% CI 2-sided [-0.89 to -0.41], Standard Error of Mean 0.1223

15. Secondary Outcome: Change From Baseline at Week 14 in Subjective Sleep Questionnaire (SSQ) - Subjective Total Sleep Time (sTST)
Description: The Subjective Sleep Questionnaire (SSQ) was included in the participant's diary and designed to capture subjective evaluation of sleep behavior in participants with disrupted sleep. It was administered to each participant approximately 30 - 60 minutes after arising each day in the morning. The Subjective Total Sleep Time (sTST) parameter subjectively estimated the total amount of time the participant was asleep after lights out until final awakening. Baseline was defined as the mean of last 7 SSQ diary entries up to and including Day 1.
Time Frame: Baseline, Week 14
Population: The Full Analysis Set (FAS) was defined as all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Minutes
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 127 | 121
Minutes | 24.63 (5.851) | 17.23 (5.958)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.3388, Mixed-effects model repeated measures — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 7.396, 95% CI 2-sided [-7.76 to 22.55], Standard Error of Mean 7.7309

16. Secondary Outcome: Change From Baseline at Week 14 in Subjective Sleep Questionnaire (SSQ) - Sleep Quality
Description: The Subjective Sleep Questionnaire (SSQ) was included in the participant's diary and designed to capture subjective evaluation of sleep behavior in participants with disrupted sleep. It was administered to each participant approximately 30 - 60 minutes after arising each day in the morning. The Sleep Quality parameter subjectively rated the quality of sleep during the past night by selecting a number between 0 (very poor) and 10 (excellent). Baseline was defined as the mean of last 7 SSQ diary entries up to and including Day 1.
Time Frame: Baseline, Week 14
Population: The Full Analysis Set (FAS) was defined as all randomized participants who received at least 1 dose of study medication.
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 127 | 123
Units on a scale | 1.59 (0.166) | 0.82 (0.169)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0003, Mixed-effects model repeated measures — [p-value comment as in outcome 1, analysis 1]; Mean Difference (Final Values) = 0.765, 95% CI 2-sided [0.35 to 1.18], Standard Error of Mean 0.2115

17. Secondary Outcome: Change From Baseline in Multidimensional Assessment of Fatigue (MAF) Score at Week 14
Description: The Multidimensional Assessment of Fatigue (MAF) scale was a self-administered survey that yielded a Global Fatigue Index by assessing the participant's level of fatigue and the degree to which fatigue interferes with activities of daily living. It contained 16 items and measured 4 dimensions of fatigue: severity (2 items), distress (1 item), degree of interference in activities of daily living (11 items), and timing (2 items). Index range was 1 to 50 and higher scores reflected greater impairment.
Time Frame: Baseline, Week 14
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 166 | 161
Units on a scale | -4.09 (0.676) | -3.25 (0.681)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.3186, ANCOVA — From the analysis of covariate (ANCOVA) with treatment and pooled center as factors, and baseline value as covariate; Mean Difference (Final Values) = -0.840, 95% CI 2-sided [-2.50 to 0.82], Standard Error of Mean 0.8414

18. Secondary Outcome: Change From Baseline at Week 14 in Short-Form 36 (SF-36) Health Survey - Mental Component Summary Score
Description: The Short-Form 36 Health Survey (SF-36) was a self-administered questionnaire that measured each of the following 8 health concepts: Physical functioning, role limitations due to physical problems, social functioning, bodily pain, mental health, role limitations due to emotional problems, vitality, and general health perception. Mental component included mental health, role limitations due to emotional problems, vitality and general health perception. Score range for mental component summary score was 0 to 100 and higher scores reflected better participant status.
Time Frame: Baseline, Week 14
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 170 | 164
Units on a scale | 2.68 (0.831) | 2.30 (0.846)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.7149, ANCOVA — From the analysis of covariate (ANCOVA) with treatment and pooled center as factors, and baseline value as covariate; Mean Difference (Final Values) = 0.380, 95% CI 2-sided [-1.67 to 2.43], Standard Error of Mean 1.0404

19. Secondary Outcome: Change From Baseline at Week 14 in Short-Form 36 (SF-36) Health Survey - Physical Component Summary Score
Description: The Short-Form 36 Health Survey (SF-36) was a self-administered questionnaire that measured each of the following 8 health concepts: Physical functioning, role limitations due to physical problems, social functioning, bodily pain, mental health, role limitations due to emotional problems, vitality, and general health perception. Physical component included physical functioning, role limitations due to physical problems, social functioning and bodily pain. Score range for physical component summary score was 0 to 100 and higher scores reflected better participant status.
Time Frame: Baseline, Week 14
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 170 | 164
Units on a scale | 4.44 (0.538) | 3.66 (0.548)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.2442, ANCOVA — From the analysis of covariate (ANCOVA) with treatment and pooled center as factors, and baseline value as covariate; Mean Difference (Final Values) = 0.785, 95% CI 2-sided [-0.54 to 2.11], Standard Error of Mean 0.6730

20. Secondary Outcome: Change From Baseline in Pain Visual Analog Scale (Pain VAS) Score at Week 14
Description: The Pain Visual Analog Scale (Pain VAS) was a horizontal line; 100 mm in length, self administered by the participants in order to rate pain from 0 "no pain" to 100 "worst possible pain".
Time Frame: Baseline, Week 14
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 170 | 164
Units on a scale | -17.04 (1.922) | -13.43 (1.952)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.1332, ANCOVA — From the analysis of covariate (ANCOVA) with treatment and pooled center as factors, and baseline value as covariate; Mean Difference (Final Values) = -3.616, 95% CI 2-sided [-8.34 to 1.11], Standard Error of Mean 2.4019

21. Secondary Outcome: Change From Baseline at Week 14 in Hospital Anxiety and Depression Scale (HADS) - Anxiety Subscale Score
Description: The Hospital Anxiety and Depression Scale (HADS) was a self-reported 14-item instrument that consisted of two 7-item subscales that measure the presence and severity of anxiety and depression. For each subscale, score range was 0 to 21, with higher scores indicating greater impairment.
Time Frame: Baseline, Week 14
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 170 | 164
Units on a scale | -1.03 (0.287) | -0.65 (0.292)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.2934, ANCOVA — From the analysis of covariate (ANCOVA) with treatment and pooled center as factors, and baseline value as covariate; Mean Difference (Final Values) = -0.378, 95% CI [-1.09 to 0.33], Standard Error of Mean 0.3595

22. Secondary Outcome: Change From Baseline at Week 14 in Hospital Anxiety and Depression Scale (HADS) - Depression Subscale Score
Description: The Hospital Anxiety and Depression Scale (HADS) was a self-reported 14-item instrument that consisted of two 7-item subscales that measure the presence and severity of anxiety and depression. For each subscale, range was 0 to 21, with higher scores indicating greater impairment.
Time Frame: Baseline, Week 14
Population: as for outcome 3
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 170 | 164
Units on a scale | -1.11 (0.290) | -0.28 (0.294)
Statistical Analysis 1: Comparison: Pregabalin vs Placebo; Test type: Superiority or Other; p = 0.0226, ANCOVA — From the analysis of covariate (ANCOVA) with treatment and pooled center as factors, and baseline value as covariate; Mean Difference (Final Values) = -0.830, 95% CI 2-sided [-1.54 to -0.12], Standard Error of Mean 0.3621

23. Secondary Outcome: Number of Participants With Treatment-Emergent Adverse Events (TEAEs), Serious Adverse Events (SAEs) and Discontinuation Due to AEs
Description: An adverse event (AE) was any untoward medical occurrence in a clinical investigation participant administered a product or medical device. A Serious adverse event (SAE) was any untoward medical occurrence at any dose that resulted in death; was life-threatening (immediate risk of death); required inpatient hospitalization or prolongation of existing hospitalization; persistent or significant disability (substantial disruption of the ability to conduct normal life functions); congenital anomaly/birth defect. Treatment-emergent AEs (TEAEs) were events between first dose of study drug and up to follow-up visit (Study Day 105) that were absent before treatment or that worsened after treatment. AEs included both SAEs and non-SAEs.
Time Frame: Baseline to Follow up (Day 105)
Population: The Safety Analysis Set was defined as all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Participants
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 170 | 164
Participants
  AEs | 119 | 103
  SAEs | 0 | 9
  Discontinuation due to AEs | 22 | 11

24. Secondary Outcome: Number of Treatment-Emergent Adverse Events (TEAEs) Categorized by Severity
Description: A mild Adverse Event (AE) was an AE that did not interfere with participant's usual function. A moderate AE was an AE that interfered participant's usual function to some extent. A severe AE was an AE that interfered significantly with participant's usual function.
Time Frame: Baseline to Follow up (Day 105)
Population: The Safety Analysis Set was defined as all randomized participants who received at least 1 dose of study medication.
Measure: Number; unit: Events
Arm/Group | Pregabalin | Placebo
Number analyzed (Participants) | 170 | 164
Events
  Mild AEs | 183 | 162
  Moderate AEs | 52 | 30
  Severe AEs | 38 | 25

ADVERSE EVENTS:
Time Frame: Baseline to Follow up (Day 105)
Arm/Group | Pregabalin | Placebo
Serious Adverse Events (participants affected / at risk) | 0/170 | 9/164
Other Adverse Events (participants affected / at risk) | 88/170 | 47/164
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=170) | Placebo (N=164)
Atrial tachycardia (Cardiac disorders) | 0 | 1
Goitre (Endocrine disorders) | 0 | 1
Bile duct stone (Hepatobiliary disorders) | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 1
Fibromyalgia (Musculoskeletal and connective tissue disorders) | 0 | 1
Cerebral haemangioma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Cerebral haemorrhage (Nervous system disorders) | 0 | 1
Vaginal haemorrhage (Reproductive system and breast disorders) | 0 | 1
Nasal obstruction (Respiratory, thoracic and mediastinal disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Pregabalin (N=170) | Placebo (N=164)
Upper respiratory tract infection (Infections and infestations) | 10 | 7
Dizziness (Nervous system disorders) | 71 | 30
Headache (Nervous system disorders) | 10 | 10
Somnolence (Nervous system disorders) | 30 | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.